CLINICAL TRIAL: NCT02722239
Title: An Open-label, Randomized, Crossover Study of Comparative Pharmacokinetics and Bioequivalence of Dapagliflozin + Metformin Modified Release Film-coated Tablets, 10 mg + 1000 mg (AstraZeneca AB, Sweden) Versus the Combined Use of Forxiga™ (Dapagliflozin), Film-coated Tablets, 10 mg (Bristol Myers Squibb Company, USA) and Two Glucophage® Long (Metformin), ER Tablets, 500 mg (Merck Santé S.A.S., France), Co-administered to Healthy Volunteers Under Standard Fed Conditions
Brief Title: An Open-label, Randomized, Crossover Study of Comparative Pharmacokinetics and Bioequivalence of Dapagliflozin + Metformin, 10 mg + 1000 mg Versus the Combined Use of Forxiga™, 10 mg and Two Glucophage® Long, ER Tablets, 500 mg Co-administered to Healthy Volunteers Under Standard Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Biocard (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1691C00012; D1691C00012 (Other: AstraZeneca)
Record Dates: First submitted 2016-03-15; First posted 2016-03-29 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Xigduo;; bioequivalence;; crossover;; Russia
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T/R (Experimental): Test product (T): a single oral dose of modified release fixed dose combination film-coated tablet consisting of 10 mg dapagliflozin IR and 1000 mg metformin hydrochloride extended release. Volunteers enrolled to group 1, on the first study period will take the study test product (Т), and on the second study period after wash out period of 7 days the volunteers will be given the Reference product (R)
  Interventions: Drug: Xigduo XR; Drug: Metformin ER (Glucophage® long); Drug: Dapagliflozin (Forxiga)
- R/T (Experimental): Reference product (R): co-administration of a single oral dose of 10 mg dapagliflozin film-coated tablet (Forxiga™) and two tablets 500 mg metformin hydrochloride extended release tablets (Glucophage® long). Volunteers from group 2 will be administered with the study drug in reverse order. It means that group 1 will take the study products in sequence T-R and group 2 in the sequence R-T.
  Interventions: Drug: Xigduo XR; Drug: Metformin ER (Glucophage® long); Drug: Dapagliflozin (Forxiga)

INTERVENTIONS:
Drug: Xigduo XR — a single oral dose of modified release fixed dose combination film-coated tablet consisting of 10 mg dapagliflozin IR and 1000 mg metformin hydrochloride extended release
Drug: Metformin ER (Glucophage® long) — co-administration of a single oral dose of 10 mg dapagliflozin film-coated tablet (Forxiga™) and two tablets 500 mg metformin hydrochloride extended release tablets (Glucophage® long).
Drug: Dapagliflozin (Forxiga) — co-administration of a single oral dose of 10 mg dapagliflozin film-coated tablet (Forxiga™) and two tablets 500 mg metformin hydrochloride extended release tablets (Glucophage® long).

SUMMARY:
The aim of this study is to demonstrate bioequivalence of fixed dose combination Dapagliflozin + Metformin modified -release, film-coated tablets, 10 mg + 1000 mg, (AstraZeneca AB, Sweden) versus Forxiga™ (Dapagliflozin), film-coated tablets, 10 mg (Bristol Myers Squibb Company, USA) and Glucophage® long (Metformin), ER tablets, 1000 mg (2 x 500 mg) (Merck Santé S.A.S., France) which are already registered in the Russian Federation.

DETAILED DESCRIPTION:
Randomised open-label crossover comparative, single center, two periods, clinical study of investigational drug and reference drugs bioequivalence evaluation with a single administration of the study drug (1 modified - release film-coated tablets of Dapagliflozin + Metformin or 1 film-coated tablets of Forxiga™ + 2 tablets ER of Glucophage® long) under fed condition in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. The volunteer is able to understand the requirements of the study, to sign the informed consent form, and agrees with all the restrictions imposed in the course of the study;
2. Male and female subjects aged 18-45, inclusive;
3. Caucasian race;
4. Body-mass index (BMI) within the range dated 18.5 to 30 kg/m2;
5. Verified diagnosis "healthy" as confirmed by the results of standard clinical, laboratory, and instrumental evaluations;
6. A negative pregnancy test at the Screening Visit for female subjects of childbearing potential.

   Postmenopausal (no menses for at least 1 year) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) females are exempted from the requirement. In case of using hormonal contraceptives, these should be withdrawn at least 2 months before the study;
7. Volunteers' with preserved reproductive potential agree to use adequate contraception throughout the study and for 30 days thereafter

Exclusion Criteria:

1. Known hypersensitivity or intolerance to dapagliflozin or metformin or any other excipient of the study drugs;
2. History of allergy to Na+ glucose co-transport inhibitor;
3. Complicated allergic history including food intolerance;
4. Lactose intolerance, lactase deficiency, glucose-galactose malabsorption;
5. Chronic diseases of the cardiovascular, bronchopulmonary, nervous, endocrine, or musculoskeletal systems, as well as diseases of the gastrointestinal tract, liver, kidneys, blood, immune system, mental disorders;
6. Deviations from the normal parameters in clinical blood count analysis, biochemical blood analysis, urinalysis; vital signs;
7. Mental, physical and other reasons that do not allow the subjects according to investigator's opinion to assess their behavior adequately, to follow correctly the requirements of the clinical study protocol and to assess the expected risks and possible discomfort;
8. Organic brain damage, history of increased seizure activity;
9. Changes on ECG (clinically significant);
10. Systolic blood pressure (AD) measured in a sitting position, less than 100 mmHg or above 130 mmHg and / or diastolic blood pressure below 70 mm Hg or above 90 mmHg at screening or any time during the study;
11. Heart rate less than 60 or more than 80 beats per minute at screening or prior to administration of the drug in each period of the study;
12. Scheduled radioisotope or radiological examinations using iodinated contrast agents during < 2 days before dosing;
13. Rare hereditary diseases manifestating with fructose or sorbitol intolerance;
14. Gastrointestinal tract surgery (except appendectomy);
15. Acute infectious diseases less than 4 weeks before the start of the study;
16. Regular medication (including dietary supplements and combination herbal medicinal products) and vitamins intake within 2 weeks (or 6 half-lives, whichever is longer) prior inclusion into the study and subject does not give agreement to refuse from this medication until the end of study;
17. Administration of the medicines that have a significant effect on circulatory dynamics, liver function, etc. (barbiturates, omeprazol, zimetidin etc.) less than 30 days before the start of the study;
18. Blood donation (450 ml and more of blood or plasma) less than 2 months before the start of the study;
19. Participation in another clinical study within 3 months before the start of the study;
20. Alcohol intake > 10 units of alcohol per week (1 unit of alcohol - 500 ml of beer, 200 ml of dry wine or 50 ml of strong alcoholic beverages) or history of alcohol abuse, narcomania or other drug abuse.
21. Use of alcohol and/or caffeinated and xanthine containing substances (for example, coffee, tea, colas, energetic drinks), chocolate as well as citrus fruits and cranberry (including juices, fruit drinks, etc.) 72 hours prior and throughout the study.
22. Smoker (>10 cigarettes per day) and/or inability to refrain from smoking on Period I and Period II
23. Special diets (e.g. vegetarians or hypocaloric diet [ less than 1000 cal/day]) or lifestyle (including night work and extreme physical activities, such as sports or weight lifting), which may impede the study conduction and monitoring;
24. Positive screening blood test for hepatitis B surface antigen (HBsAg), hepatitis C (HCV) antibody, human immunodeficiency virus (HIV-1or HIV-2 antibodies) and / or syphilis (RW);
25. A positive drug urine screening (cocaine, opiates, cannabis, barbiturates, amphetamines);
26. A positive alcohol breath test;
27. Dehydration due to diarrhea, vomiting or another cause during the last 24 hours before the start of the study;
28. There is any concern by the investigator regarding the safe participation of the subject in the study or for any other reason; the investigator considers the subject ineligible for the study.
29. Breast-feeding period;
30. For women - Use of hormonal contraceptives for 2 months before the study start;
31. Female volunteers with childbearing potential, having unprotected sexual intercourse with any unsterilized male partner (i.e., a man that is not sterilized by vasectomy for at least 6 months) for 30 days before receiving study medication.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Moscow, Russia

REFERENCES:
- [Derived] Khomitskaya Y, Tikhonova N, Gudkov K, Erofeeva S, Holmes V, Dayton B, Davies N, Boulton DW, Tang W. Bioequivalence of Dapagliflozin/Metformin Extended-release Fixed-combination Drug Product and Single-component Dapagliflozin and Metformin Extended-release Tablets in Healthy Russian Subjects. Clin Ther. 2018 Apr;40(4):550-561.e3. doi: 10.1016/j.clinthera.2018.02.006. Epub 2018 Mar 14. PMID 29548719

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from one medical clinic located in Moscow, Russia in March and April 2016.
Pre-assignment Details: 46 subjects were screened, 40 randomized (2 did not meet inclusion criteria and 4 were back-up volunteers).
Groups:
- T Drug First / Then Drug R: Test product (T): a single oral dose of modified release fixed dose combination film-coated tablet consisting of 10 mg dapagliflozin IR and 1000 mg metformin hydrochloride extended release. Volunteers enrolled to group 1, on the first study period took the study test product (Т), and on the second study period after wash out period of 7 days the volunteers were given the Reference product (R)
- R Drug First / Then Drug T: Reference product (R): co-administration of a single oral dose of 10 mg dapagliflozin film-coated tablet (Forxiga™) and two tablets 500 mg metformin hydrochloride extended release tablets (Glucophage® long). Volunteers from group 2 were administered with the study drug in reverse order. It means that group 1 took the study products in sequence T-R and group 2 in the sequence R-T.
Period: Overall Study
Arm/Group | T Drug First / Then Drug R | R Drug First / Then Drug T
Started | 20 | 20
First Intervention (1 Day) | 20 | 20
Washout (7 Days) | 20 | 20
Second Intervention (1 Day) | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The age range of the study healthy volunteers was 19-44 years.
Groups:
- Total: Total of all reporting groups
Arm/Group | T Drug First / Then Drug R | R Drug First / Then Drug T | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age (years): Mean ± Standard Deviation | 29.6 (7.7) | 30.8 (8.7) | 30.2 (8.1)
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0
  between 18 and 45 years (inclusive) | 20 | 20 | 40
  >45 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax).
Time Frame: Blood sampling 0 h, 30 min, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours and 72 hours after the dosing. Time interval for sampling is provided with pharmacokinetic characteristics of the product.
Measure: Mean (Standard Deviation); unit: ug/ml
Groups:
- Test Product (T): Test Product (T): a single oral dose of modified release fixed dose combination film-coated tablet consisting of 10 mg dapagliflozin IR and 1000 mg metformin hydrochloride extended release.
- Reference Product (R): Reference product (R): co-administration of a single oral dose of 10 mg dapagliflozin film-coated tablet (Forxiga™) and two tablets 500 mg metformin hydrochloride extended release tablets (Glucophage® long).
Arm/Group | Test Product (T) | Reference Product (R)
Number analyzed (Participants) | 40 | 40
ug/ml
  Dapagliflozin Cmax [ug/ml]: Mean (± SD) | 90.883 (25.302) | 95.975 (25.135)
  Metformin Cmax [ug/ml]: Mean (± SD) | 1030.83 (258.910) | 986.93 (255.277)

2. Primary Outcome: Area Under the "Concentration - Time" Curve (AUC0-t)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/mL*h
Arm/Group | Test Product (T) | Reference Product (R)
Number analyzed (Participants) | 40 | 40
ug/mL*h
  Dapagliflozin AUC0-t [ug/mL*h]: Mean (± SD) | 505.964 (130.420) | 511.293 (127.715)
  Metformin AUC0-t [ug/mL*h]: Mean (± SD) | 8858.52 (2998.49) | 9286.92 (3222.38)

3. Primary Outcome: Area Under the "Concentration - Time" Curve (AUC0-∞)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/mL*h
Arm/Group | Test Product (T) | Reference Product (R)
Number analyzed (Participants) | 40 | 40
ug/mL*h
  Dapagliflozin AUC0-∞ [ug/mL*h]: Mean (± SD) | 521.295 (136.036) | 532.556 (144.768)
  Metformin AUC0-∞ [ug/mL*h]: Mean (± SD) | 9408.51 (3373.65) | 9612.23 (3440.33)

4. Primary Outcome: Bioequivalence Consideration: 90% Confidence Intervals for the Test:Reference Geometric Least Squares Mean Ratios
Description: The drugs are considered bioequivalent if the 90% confidence intervals for the Test : Reference products geometric least squares mean ratios of AUC, Cmax и Cmax/AUC parameters are in the range of 80% - 125%.
Time Frame: as for outcome 1
Population: The Arms/Groups are combined because the main study goal was to compare the bioequivalence of the study drug and the reference drug which were intaken by all volunteers regardless of the group.
Measure: Least Squares Mean (90% Confidence Interval); unit: Geometric least squares mean ratio (%)
Groups:
- T Drug vs R Drug: Ratio of Test product (a single oral dose of modified release fixed dose combination film-coated tablet consisting of 10 mg dapagliflozin IR and 1000 mg metformin hydrochloride extended release) and Reference product (co-administration of a single oral dose of 10 mg dapagliflozin film-coated tablet (Forxiga™) and two tablets 500 mg metformin hydrochloride extended release tablets (Glucophage® long)).
Arm/Group | T Drug vs R Drug
Number analyzed (Participants) | 40
Geometric least squares mean ratio (%)
  Dapagliflozin AUC0-t % | 99.0829 [95.943 to 102.326]
  Dapagliflozin Cmax % | 94.7712 [87.887 to 102.194]
  Dapagliflozin Cmax/AUC0-t % | 95.6484 [89.102 to 102.675]
  Metformin AUC0-t % | 95.9105 [89.492 to 102.79]
  Metformin Cmax % | 104.3772 [98.492 to 110.614]
  Metformin Cmax/AUC0-t % | 108.8277 [101.607 to 116.561]

5. Primary Outcome: Adverse Events
Description: Adverse events data for Dapagliflozin + Metformin, modified-release film-coated tablets, 10 mg + 1000 mg (AstraZeneca AB, Sweden) and for co-administered Forxiga™ (Dapagliflozin), film-coated tablets, 10 mg, (Bristol Myers Squibb Company, USA) and Glucophage® long (Metformin), XR tablets, 500 mg/2 tablets (Merck Santé S.A.S, France)
Time Frame: AE information will be collected from the time of the first dosing to the last study procedure made in the hospital, approximately 1 month
Measure: Number; unit: adverse event
Arm/Group | Test Product (T) | Reference Product (R)
Number analyzed (Participants) | 40 | 40
adverse event | 34 | 31

ADVERSE EVENTS:
Time Frame: 1 month
Description: According to the local regulatory authorities request any (even clinically insignificant) laboratory abnormalities have been interpreted as adverse event.
Arm/Group | Test Product (T) | Reference Product (R)
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 20/40 | 19/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (T) (N=40) | Reference Product (R) (N=40)
Glucose urine present (Investigations) | 13 (13) | 9 (9) — The events were associated with dapagliflozin mechanism of action.
Haematocrit increased in hematology (Investigations) | 0 (0) | 2 (2)
Specific gravity urine decreased (Investigations) | 5 (5) | 8 (8) — The events were associated with dapagliflozin mechanism of action.
pH urine decreased (Investigations) | 15 (15) | 10 (10) — The events were associated with dapagliflozin mechanism of action.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI signed the Protocol and agreed to conform fully to the Protocol requirements. According to the Protocol the PI should inform the Sponsor in writing beforehand and provide the sponsor with all manuscripts or abstracts before submitting them to the editorial office or scientific expert board, and obtain a written permission from the Sponsor. The period is not mentioned.